CLINICAL TRIAL: NCT00489632
Title: Children's Resiliency, Adjustment, and Coping: Cancer-Related, Family Context, and Within-Child Factors
Brief Title: Children's Resiliency, Adjustment, and Coping
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2005-0628
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Leukemia
Keywords: Leukemia; Pediatrics; Cancer; Coping; Caregiver; Questionnaire; Children; Resiliency; Adjustment; Illness-related factors
MeSH Terms: conditions — Leukemia; Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Questionnaire: Children with leukemia and their families/caregivers.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaires administered to pediatric patients and their parent(s) or caregiver(s).
  Other Names: Survey

SUMMARY:
Overall Objective:

The overall objective of this cross-sectional psychosocial study is to examine illness-related factors, family context factors, and child resiliency as predictors or correlates of child adjustment to leukemia treatment.

Primary Objective 1:

1(a): To examine illness-related factors (i.e., child's health and physical functioning and severity of the child's illness) as predictors of child psychological adjustment to leukemia.

1(b): To examine relapse status as a grouping variable affecting child psychological adjustment to leukemia.

1(c): To examine stage of treatment as a grouping variable affecting child psychological adjustment to leukemia.

Primary Objective 2:

-To examine family context factors (i.e., family psychosocial risk and parental emotional distress) as correlates of child psychosocial adjustment to leukemia treatment.

Primary Objective 3:

-To examine child resiliency as a predictor of child psychological adjustment to leukemia treatment.

Secondary Objectives:

* One secondary objective of the study is to examine parental distress as a moderator affecting parental report of child adjustment to leukemia as compared to the child's self-report of adjustment.
* Another secondary objective of the study is to develop a model by which the relative contribution of each predictor variable (as determined by analyses of primary objectives) as well as their interrelatedness can be understood in relation to child psychosocial adjustment.
* A third secondary objective of the study is to examine demographic variables as covariates in the main analyses. These variables include: age, grade, site, gender, ethnicity, type of leukemia, staging, time spent in treatment, age at diagnosis, and whether the child is undergoing standard or experimental treatment.

DETAILED DESCRIPTION:
Parental Consent/Child Assent for Child Participants:

If you choose to take part in this study, you will be asked to complete a total of 2 or 3 questionnaires (depending on your age). Each questionnaire will be completed only once.

If you are between 6-7 years old, you will be given 2 questionnaires asking you about your physical health and illness, and your personal strengths. These questionnaires will take you about 30-45 minutes to finish. If you are between 8-18 years old, you will be given 3 questionnaires that will ask you about your physical health and illness, your personal strengths, and your emotional adjustment to the disease. These 3 questionnaires will take you about 30-45 minutes in total to finish. A research assistant will help you with the questionnaires, if you need help.

If you are given the questionnaires while you are at the hospital and you cannot complete them before you leave, you will be given a stamped envelope to mail the forms back to the study staff.

After your questionnaires are finished, a member of the research team might look at your medical chart if they need more information about your treatment or the status of the disease.

Parent Participants:

If you choose to take part in this study, you will be asked to complete a total of 5 questionnaires. These questionnaires ask information about your child's emotional adjustment to the disease, your child's physical health and illness, your child's personal strengths, your emotional distress, and the overall functioning of your family. Each questionnaire will be completed only once. It will take about 45-60 minutes to complete all 5 questionnaires.

Medical Staff Participants:

If you choose to take part in this study, you will be asked to complete a questionnaire that asks for information about the patient's illness. It will take about 3-5 minutes to complete this one-time survey.

All Groups:

This is an investigational study. About 220 people (100 children, 100 parents, and 20 medical staff) will take part in this multicenter study. About 130 will be enrolled at M. D. Anderson (60 children, 60 parents, and 10 medical staff members).

ELIGIBILITY:
Inclusion Criteria:

* Child who is 6 to 18 years of age or the parent or clinician of a child 6 to 18 years of age.
* The child has a diagnosis of any type of leukemia
* Child and at least one parent or non-parent caregiver must speak and read either English or Spanish well enough to complete questionnaires with some reading assistance from the researcher.
* Child is currently receiving chemotherapy treatment

Exclusion Criteria:

* If the child is currently in a medical crisis as determined by his/her primary physician (e.g., ICU admission, hospice care), he/she will not be considered for participation.
* If the child and/or parent or non-parent caregiver is unable to comprehend the survey questions, they will be excluded from participation.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children with a diagnosis of leukemia and their parent(s) or caregiver(s).
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2006-04; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Illness-related factors as predictors of child psychological adjustment to leukemia | 4 Years

CONTACTS AND LOCATIONS:
Overall Officials: Martha Askins, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - University of Minnesota Medical Center-Twin Cities, Minneapolis, Minnesota
  - UT MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org